CLINICAL TRIAL: NCT06721520
Title: Comparative Effectiveness of Intrapyloric Botulinum Toxin Injection Versus Pyloromyotomy for Pyloric Drainage During Esophagectomy: A Registry-Based, Pragmatic Randomized Noninferiority Trial
Brief Title: Effectiveness of Methods for Pyloric Drainage in esophagecTomY: Botox vs. Pyloromyotomy
Acronym: EMPTY
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Siva Raja, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 24-898
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Cancer Surgery; Esophagectomy; Delayed Gastric Emptying Following Procedure; Esophageal Diseases; Esophageal Achalasia; Pylorus Dysfunction; Esophageal Dysmotility
Keywords: Esophagectomy; Delayed gastric emptying; Delayed conduit emptying; Botox; botulinum toxin; Pyloromyotomy; Pyloric drainage
MeSH Terms: conditions — Esophageal Diseases; Esophageal Achalasia; Esophageal Motility Disorders; Gastroparesis | interventions — Botulinum Toxins, Type A; Pyloromyotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botox (Experimental): Patients will be randomized to the intrapyloric Botox injection intervention arm intraoperatively just after the pylorus is identified and just prior to the time at which pyloric drainage would occur routinely, at which point it is feasible for the surgeon to perform either intervention.
  Interventions: Biological: Botulinum Toxin A (Botox )
- Pyloromyotomy (Active Comparator): Patients will be randomized to the pyloromyotomy intervention arm intraoperatively just after the pylorus is identified and just prior to the time at which pyloric drainage would occur routinely, at which point it is feasible for the surgeon to perform either intervention.
  Interventions: Procedure: Pyloromyotomy

INTERVENTIONS:
Biological: Botulinum Toxin A (Botox ) — Patients randomized for intrapyloric Botox injection will undergo the following standard procedure: 100 units of Botox are dissolved in 10 mL normal saline. After identifying the pylorus, the 10 mL of Botox solution is injected intramuscularly at the anterior pyloric ring in 2 separate areas and in 1 area on each side of the pyloric ring.
  Arms: Botox
Procedure: Pyloromyotomy — Patients randomized for pyloromyotomy will undergo standard pyloromyotomy as follows: after identifying the pylorus, a 2-cm longitudinal incision is made with Metzenbaum or Mayo scissors on the anterior pylorus, centered on the pyloric ring. The incision extends through the serosa and muscular layers to expose the submucosa and mucosa, which is left intact. The cut muscle is spread apart until the submucosa bulges up to the level of the cut serosa. Care is taken to avoid perforation, and the surgeon confirms no mucosal perforation at the end of the procedure. If a perforation is encountered, it will be repaired primarily.
  Arms: Pyloromyotomy

SUMMARY:
The goal of this pragmatic, registry-based, randomized clinical trial is to find out if using botulinum toxin (Botox) to help drain the stomach during an esophagectomy works as well as a pyloromyotomy in patients undergoing elective esophagectomy for benign or malignant esophageal disease. Both methods are intended to prevent problems with food emptying too slowly from the stomach (delayed gastric emptying), which can cause discomfort after surgery. The main question it aims to answer is:

Is intrapyloric Botox injection as a drainage procedure during esophagectomy non-inferior in preventing symptoms of delayed gastric emptying at 6 months postoperatively compared to pyloromyotomy?

Researchers will compare intrapyloric Botox injection to pyloromyotomy to see if Botox is non-inferior to pyloromyotomy in easing symptoms of delayed gastric emptying.

Participants will:

Be randomized to one of two treatment groups-either intrapyloric Botox injection or pyloromyotomy-during their esophagectomy.

Complete surveys assessing digestive symptoms at standard postoperative follow-up intervals (3 months, 6 months, 1 year, and 2 years postoperatively).

Undergo a standard gastric emptying study at 6 months after surgery.

DETAILED DESCRIPTION:
This is a single institution, pragmatic, registry-based, prospective, single-blinded, randomized, double-arm, noninferiority clinical trial comparing outcomes of two standard-of-care alternative intraoperative methods of pyloric drainage during esophagectomy. One arm of the study will be patients receiving intervention 1, intrapyloric Botox injection (Botox Group), and the other arm will be patients receiving intervention 2, pyloromyotomy (Pyloromyotomy Group). Participants will be allocated equally to the interventions being compared (allocation ratio 1:1).

Patients randomized for intrapyloric Botox injection will undergo our standard procedure as follows: 100 units of Botox is dissolved in 10 mL normal saline. After identifying the pylorus during esophagectomy, 10 mL of the Botox solution is injected intramuscularly at the anterior pyloric ring in 2 separate areas and in 1 area on each side of the pyloric ring (total 4 areas). Patients randomized for pyloromyotomy will undergo standard pyloromyotomy through a transabdominal, anterior approach.

This study will occur at Cleveland Clinic Foundation in Cleveland, OH. Three staff surgeons will perform these operations.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergoing elective esophagectomy (thoracoabdominal, Ivor-Lewis, McKeown)
* Receiving a gastric conduit for alimentary reconstruction
* Technically able to receive either intrapyloric Botox injection or pyloromyotomy as ultimately determined intraoperatively
* Willing and able to provide informed consent
* Willing and able to participate in long-term follow up including study visits and surveys

Exclusion Criteria:

* Undergoing emergent esophagectomy (e.g., for esophageal perforation)
* Patients with underlying neuromuscular disease as Botox would be contraindicated (amyotrophic lateral sclerosis, myasthenia gravis, muscular dystrophies, Lambert-Eaton syndrome)
* Patients undergoing left thoracoabdominal without left cervical neck incision (i.e., Sweet esophagectomy) - excluded due to the extent of gastric resection
* Pregnancy
* Allergy or hypersensitivity to botulinum toxin
* Cannot feasibly receive both pyloric interventions as determined intraoperatively (e.g., patients with central obesity undergoing thoracoabdominal esophagectomy makes for a technically difficult pyloromyotomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Gastroparesis Cardinal Symptom Index (GCSI) total score at 6 months postoperatively or prior to the first reintervention (which ever comes first) | 6 months postoperatively or prior to the first pyloric reintervention to treat symptoms of delayed gastric emptying postoperatively (whichever comes first)
  The GCSI is a validated 9-item instrument used to quantify severity of symptoms associated with delayed gastric emptying. The GCSI is based on three subscales, which measure cardinal symptoms related to delayed gastric emptying: postprandial fullness/early satiety (4 items), nausea/vomiting (3 items), and bloating (2 items). A 6-point Likert-type response scale, ranging from 0 (none) to 5 (very severe) is used for rating the severity of each symptom item, with a recall period of 2 weeks. Subscale scores are calculated by averaging across the item scores within each subscale. The range of subscale scores is 0 to 5, where higher scores reflect perception of worse symptom severity. The GCSI total score is constructed as the average of the three symptom subscales scores. GCSI. GSCI scores will be obtained preoperatively and at 3-month, 6-month, 1-year, and 2-year follow up, with 6 months as the specific time point for our primary endpoint.

SECONDARY OUTCOMES:
Complications in the immediate post-operative period (within 30 days post-operatively) | 30 days postoperatively or until discharge from the index hospitalization (whichever duration is greater)
  Perioperative complications include gastroesophageal anastomotic leaks, pyloric leaks, aspiration, pneumonia, respiratory failure, cardiac arrhythmia, myocardial infarction, cardiac failure, mortality, and readmission within 30 days for nausea/vomiting or pneumonia. These outcomes are routinely recorded by trained registry personnel at our institution as part of national quality reporting requirements.
Gastric emptying at 6 months postoperatively, measured by gastric emptying scintigraphy study (GES) | 6 months postoperatively
  At 6 months postoperatively, a 4-hour solid-phase GES, considered the gold standard for assessing gastric motility, will be obtained as per our institute's standard of care and interpreted by Cleveland Clinic radiologists. The study consists of administering a low-fat, egg-white meal containing technetium-99m sulfur colloid labeled egg albumin. Gastric retention of the egg meal is measured at baseline and at 1, 2, and 4 hours after consumption and the results are reported as a retained percentage. Also included in the radiology report is the half-emptying time, or the time the stomach requires to empty 50% of the ingested radiolabeled test solid meal, which is commonly used to assess gastric emptying in post-esophagectomy studies. Due to the non-linear nature of gastric emptying, we will also use the percentage of food retained at 4 hours as an additional measure, which has been a marker of delayed gastric emptying in previous research.
Cleveland Clinic Esophageal Questionnaire (CEQ) domain scores at 6-months postoperatively or prior to the first reintervention (whichever comes first) | 6 months postoperatively or prior to the first pyloric reintervention to treat symptoms of delayed gastric emptying postoperatively (whichever comes first)
  The impact of symptom severity on patient quality of life (QoL) will be assessed by Cleveland Clinic Esophageal Questionnaire (CEQ) raw domain scores. The CEQ is a validated patient-reported outcome measure that allows for quantification of esophageal symptoms and their impact on the patient's quality of life. The CEQ is comprised of 34 items divided into 6 domains: dysphagia (7 items), eating (7 items), pain (5 items), reflux/regurgitation (5 items), dyspepsia (4 items), and dumping (6 items). Each item is accompanied by a question regarding frequency of symptoms, with a 6-point Likert-type response option ranging from 1 (never) to 6 (several times a day) and a question regarding the symptom's impact on quality of life, with a 5-point Likert-type response option ranging from 1 (not at all) to 5 (a lot). We will obtain the raw scores across each domain at baseline preoperatively and at 3-months, 6-months, 1-year, and 2-years follow-up, per our institution's standard of care protocol.
Pyloric reinterventions by 24 months post-operatively | 24 months postoperatively
  After esophagectomy, patients reporting severe symptoms related to delayed gastric emptying, determined based upon standard clinical evaluation (i.e., patients with a moderate or large amount of retained food on routine, post-operative upper endoscopy after fasting for 8 hours and reporting severe regurgitation or having an aspiration pneumonia event), will be offered further endoscopic treatment of their delayed gastric emptying, per our institute's standard of care protocol. We will compare frequency of reinterventions up until 24-months postoperatively in each arm. Per our institution's protocol, all of these patients, regardless of which treatment arm they are in, initially receive endoscopic Botox injection. If their gastric emptying improves, demonstrated by improvement of GCSI score or decrease in amount of retained food on upper endoscopy, and they do not have symptoms of dumping syndrome, they are then offered gastric per-oral endoscopic pyloromyotomy (G-POEM).

CONTACTS AND LOCATIONS:
Overall Officials: Siva Raja, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan OA, Manners J, Rengarajan A, Dunning J. Does pyloroplasty following esophagectomy improve early clinical outcomes? Interact Cardiovasc Thorac Surg. 2007 Apr;6(2):247-50. doi: 10.1510/icvts.2006.149500. Epub 2006 Dec 18. PMID 17669829
- [Background] Urschel JD, Blewett CJ, Young JE, Miller JD, Bennett WF. Pyloric drainage (pyloroplasty) or no drainage in gastric reconstruction after esophagectomy: a meta-analysis of randomized controlled trials. Dig Surg. 2002;19(3):160-4. doi: 10.1159/000064206. PMID 12119515
- [Background] Fok M, Cheng SW, Wong J. Pyloroplasty versus no drainage in gastric replacement of the esophagus. Am J Surg. 1991 Nov;162(5):447-52. doi: 10.1016/0002-9610(91)90258-f. PMID 1951907
- [Background] Deng B, Tan QY, Jiang YG, Zhao YP, Zhou JH, Chen GC, Wang RW. Prevention of early delayed gastric emptying after high-level esophagogastrostomy by "pyloric digital fracture". World J Surg. 2010 Dec;34(12):2837-43. doi: 10.1007/s00268-010-0766-z. PMID 20734044
- [Background] Arya S, Markar SR, Karthikesalingam A, Hanna GB. The impact of pyloric drainage on clinical outcome following esophagectomy: a systematic review. Dis Esophagus. 2015 May-Jun;28(4):326-35. doi: 10.1111/dote.12191. Epub 2014 Feb 24. PMID 24612489
- [Background] Sutcliffe RP, Forshaw MJ, Tandon R, Rohatgi A, Strauss DC, Botha AJ, Mason RC. Anastomotic strictures and delayed gastric emptying after esophagectomy: incidence, risk factors and management. Dis Esophagus. 2008;21(8):712-7. doi: 10.1111/j.1442-2050.2008.00865.x. Epub 2008 Oct 1. PMID 18847448
- [Background] Benedix F, Willems T, Kropf S, Schubert D, Stubs P, Wolff S. Risk factors for delayed gastric emptying after esophagectomy. Langenbecks Arch Surg. 2017 May;402(3):547-554. doi: 10.1007/s00423-017-1576-7. Epub 2017 Mar 21. PMID 28324171
- [Background] Hajibandeh S, Hajibandeh S, McKenna M, Jones W, Healy P, Witherspoon J, Blackshaw G, Lewis W, Foliaki A, Abdelrahman T. Effect of intraoperative botulinum toxin injection on delayed gastric emptying and need for endoscopic pyloric intervention following esophagectomy: a systematic review, meta-analysis, and meta-regression analysis. Dis Esophagus. 2023 Oct 27;36(11):doad053. doi: 10.1093/dote/doad053. PMID 37539558
- [Background] Konradsson M, Nilsson M. Delayed emptying of the gastric conduit after esophagectomy. J Thorac Dis. 2019 Apr;11(Suppl 5):S835-S844. doi: 10.21037/jtd.2018.11.80. PMID 31080667
- [Background] Tcherniak A, Kashtan DH, Melzer E. Successful treatment of gastroparesis following total esophagectomy using botulinum toxin. Endoscopy. 2006 Feb;38(2):196. doi: 10.1055/s-2006-925148. No abstract available. PMID 16479431
- [Background] Stewart CL, Wilson L, Hamm A, Bartsch C, Boniface M, Gleisner A, Mitchell JD, Weyant MJ, Meguid R, Gajdos C, Edil BH, McCarter M. Is Chemical Pyloroplasty Necessary for Minimally Invasive Esophagectomy? Ann Surg Oncol. 2017 May;24(5):1414-1418. doi: 10.1245/s10434-016-5742-x. Epub 2017 Jan 5. PMID 28058546
- [Background] Giugliano DN, Berger AC, Meidl H, Pucci MJ, Rosato EL, Keith SW, Evans NR, Palazzo F. Do intraoperative pyloric interventions predict the need for postoperative endoscopic interventions after minimally invasive esophagectomy? Dis Esophagus. 2017 Apr 1;30(4):1-8. doi: 10.1093/dote/dow034. PMID 28375478
- [Background] Tham JC, Nixon M, Ariyarathenam AV, Humphreys L, Berrisford R, Wheatley T, Sanders G. Intraoperative pyloric botulinum toxin injection during Ivor-Lewis gastroesophagectomy to prevent delayed gastric emptying. Dis Esophagus. 2019 Jun 1;32(6):doy112. doi: 10.1093/dote/doy112. PMID 30561584
- [Background] Cerfolio RJ, Bryant AS, Canon CL, Dhawan R, Eloubeidi MA. Is botulinum toxin injection of the pylorus during Ivor Lewis [corrected] esophagogastrectomy the optimal drainage strategy? J Thorac Cardiovasc Surg. 2009 Mar;137(3):565-72. doi: 10.1016/j.jtcvs.2008.08.049. PMID 19258066
- [Background] Martin JT, Federico JA, McKelvey AA, Kent MS, Fabian T. Prevention of delayed gastric emptying after esophagectomy: a single center's experience with botulinum toxin. Ann Thorac Surg. 2009 Jun;87(6):1708-13; discussion 1713-4. doi: 10.1016/j.athoracsur.2009.01.075. PMID 19463583
- [Background] Bagheri R, Fattahi SH, Haghi SZ, Aryana K, Aryanniya A, Akhlaghi S, Riyabi FN, Sheibani S. Botulinum toxin for prevention of delayed gastric emptying after esophagectomy. Asian Cardiovasc Thorac Ann. 2013 Dec;21(6):689-92. doi: 10.1177/0218492312468438. Epub 2013 Jul 11. PMID 24569327
- [Background] Eldaif SM, Lee R, Adams KN, Kilgo PD, Gruszynski MA, Force SD, Pickens A, Fernandez FG, Luu TD, Miller DL. Intrapyloric botulinum injection increases postoperative esophagectomy complications. Ann Thorac Surg. 2014 Jun;97(6):1959-64; discussion 1964-5. doi: 10.1016/j.athoracsur.2013.11.026. Epub 2014 May 1. PMID 24793689
- [Background] Marchese S, Qureshi YA, Hafiz SP, Dawas K, Turner P, Mughal MM, Mohammadi B. Intraoperative Pyloric Interventions during Oesophagectomy: a Multicentre Study. J Gastrointest Surg. 2018 Aug;22(8):1319-1324. doi: 10.1007/s11605-018-3759-0. Epub 2018 Apr 17. PMID 29667092
- [Background] Fuchs HF, Broderick RC, Harnsberger CR, Divo FA, Coker AM, Jacobsen GR, Sandler BJ, Bouvet M, Horgan S. Intraoperative Endoscopic Botox Injection During Total Esophagectomy Prevents the Need for Pyloromyotomy or Dilatation. J Laparoendosc Adv Surg Tech A. 2016 Jun;26(6):433-8. doi: 10.1089/lap.2015.0575. Epub 2016 Apr 4. PMID 27043862
- [Background] Kent MS, Pennathur A, Fabian T, McKelvey A, Schuchert MJ, Luketich JD, Landreneau RJ. A pilot study of botulinum toxin injection for the treatment of delayed gastric emptying following esophagectomy. Surg Endosc. 2007 May;21(5):754-7. doi: 10.1007/s00464-007-9225-9. Epub 2007 Feb 16. PMID 17458616